CLINICAL TRIAL: NCT01097304
Title: Clinical Study of Ursodeoxycholic Acid in Barrett's Patients
Brief Title: Ursodiol in Treating Patients With Barrett Esophagus and Low-Grade Dysplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2012-00450; NCI-2012-00450 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000669111; 09-0141-03 (Other: University of Arizona Health Sciences Center); UAZ08-11-01 (Other: DCP); P50CA095060 (NIH); N01CN35158 (NIH); P30CA023074 (NIH)
Record Dates: First submitted 2010-03-31; First posted 2010-04-01 (Estimated); Results first posted 2015-05-15 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-11

CONDITIONS: Barrett Esophagus; Esophageal Carcinoma
MeSH Terms: conditions — Barrett Esophagus; Esophageal Neoplasms | interventions — Ursodeoxycholic Acid

ARMS (1):
- Treatment (ursodiol) (Experimental): Patients receive ursodiol PO BID for 6 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ursodiol; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Ursodiol — Given PO
  Other Names: Actigall; Deursil; UDCA; URSO
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This pilot phase II trial studies how well ursodiol works in treating patients with Barrett esophagus or cells that look abnormal under a microscope but are not cancer (low-grade dysplasia). Chemoprevention is the use of certain drugs to keep cancer from forming. The use of ursodiol may keep cancer for forming in patients with Barrett esophagus or low-grade dysplasia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the ability of UDCA (ursodiol) treatment to reverse oxidative deoxyribonucleic acid (DNA) damage in the esophageal epithelium of subjects with Barrett's esophagus.

SECONDARY OBJECTIVES:

I. To determine the effects of UDCA treatment on gastric bile acid composition and on cell proliferation in Barrett's epithelium.

OUTLINE:

Patients receive ursodiol orally (PO) twice daily (BID) for 6 months in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up for 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Barrett's esophagus with histologically-confirmed intestinal metaplasia anywhere in the tubular esophagus either with >= 2 cm of involvement or with a minimum circumferential Barrett's esophagus (BE) length of 1 cm
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Leukocytes >= 3,000/uL
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Total bilirubin =< 2.0 mg/dL
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) =< 2 X institutional upper limit of normal (ULN)
* Creatinine =< 1X ULN
* Women of child-bearing potential (i.e., not surgically sterile or less than one year since last menstrual period) agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; women of childbearing potential must have a negative urine pregnancy test within 14 days prior to study agent administration; male subjects must agree to use adequate contraception (barrier method, abstinence, subject has had vasectomy or partner is using effective birth control or is postmenopausal)
* Ability to understand and the willingness to sign a written informed consent document
* Agree to refrain from any non-steroidal anti-inflammatory drug (NSAID) with the exception of low-dose aspirin (81 mg once daily [QD]) during the entire study period
* Agree not to take aluminum-containing antacids and anion exchange resins such as cholestyramine, colestimide or colestipol within 2 hours of taking UDCA

Exclusion Criteria:

* Barrett's esophagus with high grade dysplasia or carcinoma at enrollment
* Medical conditions which would make completing endoscopies or completing the trial difficult including but not limited to previous transient ischemic attacks or cerebral vascular disease, severe respiratory disease, severe ischemic heart disease or myocardial infarction in the previous 6 months, inflammatory bowel disease
* Participants may not be receiving any other investigational agents within 1 month of study enrollment
* Have used NSAID for more than 5 days per month within 1 month of enrollment except low dose aspirin (81 mg QD)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to UDCA
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant and breastfeeding women are excluded from this study; breastfeeding should be discontinued during treatment; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately
* Have had major upper gastrointestinal (GI) surgeries within 6 months of enrollment including, but not limited to, fundoplication, bariatric surgery, cholecystectomy
* Erosive esophagitis detected at the baseline endoscopy
* Participants who need concurrent chemotherapy, radiotherapy, or cancer-related hormonal or immunotherapy during the time of study
* Participants who have had chemotherapy, radiotherapy, or cancer-related hormonal or immunotherapy within 18 months of the baseline visit
* Current or planned use of anticoagulant drugs including, but not limited to, warfarin, heparin, low molecular weight heparin, Plavix, or Aggrenox
* Use of cyclosporine during the time of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-04; Primary Completion 2014-04 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bhaskar Banerjee, Principal Investigator — University of Arizona Health Sciences Center
Locations (4):
- United States (4):
  - Southern Arizona Veterans Affairs Health Center, Tucson, Arizona
  - Arizona Cancer Center-North Campus, Tucson, Arizona
  - University of Arizona Health Sciences Center, Tucson, Arizona
  - University of North Carolina, Chapel Hill, North Carolina

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Ursodiol): Patients receive ursodiol PO (13 to 15 mg/kg/day) BID for 6 months in the absence of disease progression or unacceptable toxicity.
  Ursodiol: Given PO
  Laboratory Biomarker Analysis: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Ursodiol)
Started | 36
Completed | 29
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Ursodiol)
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 30
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Reversal of Oxidative DNA Damage as Assessed by Changes in 8-hydroxy-2' -Deoxyguanosine (8OHdG) Immunostaining
Description: 8OHdG will be assessed by percentage of positively stained nuclear area. A paired t-test at a one-sided 0.05 significance level will be used to assess change during intervention. The observed results will be reported along with the corresponding confidence intervals.
Time Frame: Baseline to 6 months
Population: participants with fewer than 500 total nuclei in longitudinally sectioned crypts opening to the lumen were excluded from analysis
Measure: Mean (Standard Deviation); unit: % of strongly/moderately stained nuclei
Arm/Group | Treatment (Ursodiol)
Number analyzed (Participants) | 25
% of strongly/moderately stained nuclei | 1.62 (13.13)
Statistical Analysis 1: Comparison: Treatment (Ursodiol); Test type: Other; p = 0.54, t-test, 2 sided

2. Secondary Outcome: Changes in Gastric Bile Acid Composition (Change in Percent of Total Bile Acid Present as Ursodeoxycholic Acid and Its Glycine/Taurine Conjugates) Measured by Liquid Chromatography-tandem Mass Spectrometry, From Baseline to Post-intervention
Time Frame: Baseline and 6 months
Population: analysis was limited to participants with baseline and 6-month gastric fluid
Measure: Median (Inter-Quartile Range); unit: % of total bile acid
Arm/Group | Treatment (Ursodiol)
Number analyzed (Participants) | 28
% of total bile acid | 66.28 [36.29 to 77.09]
Statistical Analysis 1: Comparison: Treatment (Ursodiol); Test type: Other; p < 0.0001, signed rank test

3. Secondary Outcome: Changes in Gastric Bile Acid Composition (Change in Percent of Total Bile Acid Present as Deoxycholic Acid and Its Glycine/Taurine Conjugates) Measured by Liquid Chromatography-tandem Mass Spectrometry, From Baseline to Post-intervention
Time Frame: Baseline and 6 months
Population: analysis was limited to participants with baseline and 6-month gastric fluid
Measure: Median (Inter-Quartile Range); unit: % of total bile acid
Arm/Group | Treatment (Ursodiol)
Number analyzed (Participants) | 28
% of total bile acid | -13.31 [-46.98 to 0.4]
Statistical Analysis 1: Comparison: Treatment (Ursodiol); Test type: Other; p < 0.01, signed rank test

4. Secondary Outcome: Changes in Cell Proliferation in BE Epithelium From Baseline to Post-intervention as Assessed by Proliferation-related Ki-67 Antigen (Ki67) Immunostaining, Percentage of Positively Stained Nuclei, in BE Tissue Sections
Description: Results will be analyzed using paired t-tests. Results (mean values and changes during intervention) will be reported along with the corresponding confidence intervals.
Time Frame: Baseline and 6 months
Population: tissue slides with fewer than 500 total nuclei in longitudinally sectioned crypts opening to the lumen were excluded from analysis
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | Treatment (Ursodiol)
Number analyzed (Participants) | 29
% change | 1.36 (13.13)
Statistical Analysis 1: Comparison: Treatment (Ursodiol); Test type: Other; p = 0.48, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Treatment (Ursodiol)
Serious Adverse Events (participants affected / at risk) | 5/36
Other Adverse Events (participants affected / at risk) | 31/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Ursodiol) (N=36)
Hypotension (Cardiac disorders) | 1
Ischemia/Infarction (Cardiac disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Barrett's esophagus with at least intramucosal carcinoma (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Post surgical pain (Musculoskeletal and connective tissue disorders) | 1
CNS cerebrovascular ischemia (Nervous system disorders) | 1
Altered mental status (Nervous system disorders) | 1
Chest/Thorax pain (Cardiac disorders) | 1
Renal failure (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Ursodiol) (N=36)
hypertension (Cardiac disorders) | 2
Fatigue (General disorders) | 4
Fever (General disorders) | 2
Weight loss (Investigations) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 3
Colitis (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 10
Distention/Bloating (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 2
Heartburn (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 7
Phytobezoar (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 6
Upper airway infection (Infections and infestations) | 6
Hyponatremia (Metabolism and nutrition disorders) | 2
Dizziness (Nervous system disorders) | 6
Abdomen pain (Gastrointestinal disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3
Headache (Nervous system disorders) | 6
Joint pain (Musculoskeletal and connective tissue disorders) | 3
Stomach pain (Gastrointestinal disorders) | 3
Phlebitis (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less